CLINICAL TRIAL: NCT07363941
Title: COMPARISON OF HEMODYNAMIC AND ANAESTHETIC OUTCOMES BETWEEN HEIGHT-BASED AND CONVENTIONAL SPINAL ANAESTHETIC DOSING IN GERIATRIC PATIENTS UNDERGOING LOWER LIMB ORTHOPAEDIC SURGERIES
Brief Title: HEIGHT-BASED AND CONVENTIONAL SPINAL ANAESTHETIC DOSING IN GERIATRIC PATIENTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaheed Mohtarma Benazir Bhutto Institue of Trauma (Other)
Responsible Party: Principal Investigator, Jehanzaib Muhammad Azam, Jehanzaib Muhammad Azam, Shaheed Mohtarma Benazir Bhutto Institue of Trauma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-000210/SMBBIT/Approval/20
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Geriatric Population; Spinal Anesthesia Induced Hypotension; Spinal Anesthesia in Elderly Patients

STUDY DESIGN:
Intervention Model Description: Group A will receive 0.07 mg/cm of 0.5% Hyperbaric Bupivacaine in conjunction with 2 mg (0.5 ml) of preservative-free Dexamethasone administered intrathecally, whereas patients in Group B will be administered 12.5 mg (2.5 ml) of 0.5% Hyperbaric Bupivacaine alongside 2 mg (0.5 ml) of preservative-free Dexamethasone
Who Masked: Outcomes Assessor
Masking Description: This study is single blind, assessor is kept blind because participants are difficult to mask due to well distinguished treatment plan.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants will receive 0.07 mg/cm of 0.5% Hyperbaric Bupivacaine in conjunction with 2 mg (0.5 ml) of preservative-free Dexamethasone administered intrathecally
  Interventions: Drug: Group A : Spinal Anaesthetic Dose
- Group B (Active Comparator): Participants will recieve 12.5 mg (2.5 ml) of 0.5% Hyperbaric Bupivacaine alongside 2 mg (0.5 ml) of preservative-free Dexamethasone administered intrathecally
  Interventions: Drug: Group B : Conventional Dose

INTERVENTIONS:
Drug: Group A : Spinal Anaesthetic Dose — Participants will receive 0.07 mg/cm of 0.5% Hyperbaric Bupivacaine in conjunction with 2 mg (0.5 ml) of preservative-free Dexamethasone administered intrathecally
  Arms: Group A
Drug: Group B : Conventional Dose — Participants will receive 12.5 mg (2.5 ml) of 0.5% Hyperbaric Bupivacaine alongside 2 mg (0.5 ml) of preservative-free Dexamethasone intrathecally
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to find out whether height-based dosing of spinal anaesthesia provides better hemodynamic stability and anesthetic outcome than conventional fixed dosing in elderly patients undergoing lower limb orthopaedic surgery.The main questions this study aims to answer are:

1. Does height-based spinal anaesthetic dosing reduce the risk of hypotension and bradycardia during surgery as compared to conventional fixed dosing?
2. Does it improve anaesthetic outcomes, such as the onset and duration of sensory and motor block?

DETAILED DESCRIPTION:
Data collection would begin after the approval of ethical review committee of the institution. This investigation will encompass patients who are scheduled to undergo lower limb orthopaedic surgical procedures within the Department of Anaesthesia, SMBBIT, Karachi. Following a comprehensive description of the study and their acceptance to participate (written consent), the subject will be recruited as detailed in the inclusion criteria.

Data will be collected using a defined data collection proforma to record baseline demographics and clinical characteristics including age, height, gender, and residential status. Height will be measured in the supine position as the patients will be undergoing lower limb surgeries. The patient will be placed flat on a firm examination table or operating-room bed without a pillow, with legs extended and neutral. To accurately measure height in centimetres, a measuring tape or stadiometer will be placed along the length of the patient's body from the heel to the vertex of the head, using trained staff to ensure precise placement, and the reading will be recorded to the nearest decimal point.

The subjects will be allocated to one of two groups through a computer-generated random number sequence with concealed allocation to mitigate selection bias and safeguard the integrity of the randomization process. Allocation concealment will be accomplished by the Sequentially Numbered, Opaque, Sealed Envelope (SNOSE) method, conducted by a blinded independent researcher not involved in subject recruitment, surgical procedure, or clinical assessment. In the operating room, baseline pulse rate and mean arterial pressure will be measured before spinal anaesthesia is induced. Intravenous access will be established, and patients will be preloaded with Ringer Lactate (10 ml/kg) prior to induction of spinal anaesthesia.

Spinal anaesthesia will be provided in the sitting position, aseptically at the level of L3-4 vertebra. Group A will receive 0.07 mg/cm of 0.5% Hyperbaric Bupivacaine in conjunction with 2 mg (0.5 ml) of preservative-free Dexamethasone administered intrathecally, whereas patients in Group B will be administered 12.5 mg (2.5 ml) of 0.5% Hyperbaric Bupivacaine alongside 2 mg (0.5 ml) of preservative-free Dexamethasone. Subsequent to the administration of spinal anaesthesia, patients will be positioned in the supine orientation; sensory blockade will be evaluated utilizing the pinprick method with a blunt-tipped 23-gauge needle at the T10 dermatome level, while motor blockade will be assessed employing the Bromage scale. The specific time at which the most effective sensory and motor blockade is achieved will be documented in accordance with the established operational definition.

The hemodynamic (heart rate and mean arterial pressure) will be continuously monitored. The procedure and the principal investigator (in consultation with a faculty consultant with >5 years' experience) will mark the findings of "bradycardia" and "hypotension" based on the operational definition on the proforma. The early postoperative period will be followed in all patients in order to know sensory and motor blockade duration by operational definition, and each result will be written. The principal investigator will record collected data on a predesigned proforma. Confidentiality will be ensured along with data security measures allowing only authorized personnel access to all information. The study is produced to be directly relevant with its aims, and rigorous exclusion criteria will be used in minimizing potential biases or confounders.

Data will be entered into a secure database and analyzed using SPSS version 26. Continuous variables (including age, height, weight, BMI, heart rate, mean arterial pressure, onset of sensory block, and duration of sensory block) will be summarized as mean ± standard deviation or median with interquartile range, as appropriate. Comparisons between the two study groups will be performed using the independent sample t-test for continuous variables. Chi-square test or Fisher's exact test will be used for categorical variables, depending on expected cell counts. A p-value ≤ 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged 60 to 80 years. Either gender (male or female). Patients who are ASA physical status I-III. Individuals scheduled to undergo elective lower limb orthopaedic surgeries (e.g., fracture fixation, total knee replacement, open reduction and internal fixation).

Patients planned to receive spinal anaesthesia as the primary anaesthetic technique.

Those who provide informed written consent for participation in the study.

Exclusion Criteria:

Individuals exhibiting a stature inferior to 150 cm. Patients receiving anti-hypertensive drugs or those on beta blockers or beta-agonists.

Patients with a history of neurological disease like CVA or Parkinsonism. Patients presenting with sepsis (≥ 2 positive SIRS criteria with positive aseptically obtained blood or wound culture).

Patients with a history of coagulation disorders like haemophilia or vWD or those with a history of anti-platelet drug intake in the last 2 weeks.

Individuals possessing a documented history of hypersensitivity reactions to pharmacological agents utilized in the research.

Patients who will be diagnosed with a skin infection at the spinal needle puncture site.

Patients undergoing emergency orthopaedic procedures requiring immediate intervention

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-01-03 (Actual); Primary Completion 2026-05-03 (Estimated); Study Completion 2026-05-04 (Estimated)

PRIMARY OUTCOMES:
HYPOTENSION | Subsequent to the administration of spinal anaesthesia till the end of sensory and motor blockade
  Defined as a decrease of ≥20% in mean arterial pressure (MAP) from baseline or an absolute MAP <65 mmHg at any point during surgery, recorded using non-invasive blood pressure monitoring at five-minute intervals
BRADYCARDIA | Subsequent to the administration of spinal anaesthesia till the end of sensory and motor blockade
  It will be defined in terms of a heart rate of ≤ 60 beats/minute during surgery
ONSET OF SENSORY BLOCK | Subsequent to the administration of spinal anaesthesia till the attainment of sensory blockade
  It will be defined as the time interval (in minutes) from the completion of intrathecal injection of bupivacaine to the loss of pinprick sensation at the T10 dermatome. The assessment will be carried out using a sterile blunt 23-gauge needle at one-minute intervals until loss of sensation is confirmed.
DURATION OF SENSORY BLOCK | Subsequent to the administration of spinal anaesthesia till the end of sensory blockade
  It will be defined as the time interval (in minutes) from the onset of sensory block at the T10 dermatome (confirmed by loss of pinprick sensation) to the reappearance of sensation at the same dermatome level. The response will be assessed every 5 minutes using a sterile blunt 23-gauge needle.
ONSET OF MOTOR BLOCK | Subsequent to the administration of spinal anaesthesia till the attainment of motor blockade
  It will be defined as the time duration (in minutes) between the completion of intrathecal administration of bupivacaine until the patient develops Bromage III
DURATION OF MOTOR BLOCK | Subsequent to the administration of spinal anaesthesia till the end of motor blockade
  The duration of motor block is defined as the time duration (in minutes) from the onset of motor block (inability to move feet) until the patient regains the ability to voluntarily move both feet.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaheed Mohtarma Benazir Bhutto Institue of Trauma, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patient Confidentiality: Sharing IPD could compromise patient confidentiality and anonymity.
  Informed consent: Participants are not providing informed consent for their data to be shared and it could raise ethical concerns.

REFERENCES:
- [Background] Hasan SH. Randomized controlled trial on the effects of fixed-dose versus height-adjusted dose of hyperbaric bupivacaine used in spinal anaesthesia for cesarean section. J Nat Sc Biol Med. 2024;15(2):192-201.
- [Background] Alkonaiesy RM, Amin SM, Abdallah NM, Muhammad SI, Hassan H. Effect of height-based spinal anaesthetic dose versus conventional dose on hemodynamics in lower limb surgeries in geriatric patients: a randomized controlled trial. Anaesth Pain Intensive Care. 2023;27(4):565-72.
- [Background] Nazli B, Oguzalp H, Horasanli E, Gamli M, Dikmen B, Gogus N. The effects on sensorial block, motor block, and haemodynamics of levobupivacaine at different temperatures applied in the subarachnoid space. Biomed Res Int. 2014;2014:132687. doi: 10.1155/2014/132687. Epub 2014 Mar 18. PMID 24772412
- [Background] Messina A, La Via L, Milani A, Savi M, Calabro L, Sanfilippo F, Negri K, Castellani G, Cammarota G, Robba C, Morenghi E, Astuto M, Cecconi M. Spinal anesthesia and hypotensive events in hip fracture surgical repair in elderly patients: a meta-analysis. J Anesth Analg Crit Care. 2022 May 8;2(1):19. doi: 10.1186/s44158-022-00047-6. PMID 37386657
- [Background] Visavakul O, Leurcharusmee P, Pipanmekaporn T, Khorana J, Patumanond J, Phinyo P. Effective Dose Range of Intrathecal Isobaric Bupivacaine to Achieve T5-T10 Sensory Block Heights for Elderly and Overweight Patients: An Observational Study. Medicina (Kaunas). 2023 Mar 1;59(3):484. doi: 10.3390/medicina59030484. PMID 36984485
- [Background] Al Harbi MK, Alshaghroud SM, Aljahdali MM, Ghorab FA, Baba F, Al Dosary R, Bahadeq M. Regional anesthesia for geriatric population. Saudi J Anaesth. 2023 Oct-Dec;17(4):523-532. doi: 10.4103/sja.sja_424_23. Epub 2023 Aug 18. PMID 37779559
- [Background] Lim BG, Lee IO. Anesthetic management of geriatric patients. Korean J Anesthesiol. 2020 Feb;73(1):8-29. doi: 10.4097/kja.19391. Epub 2019 Oct 22. PMID 31636241
- [Background] Neuman MD, Feng R, Carson JL, Gaskins LJ, Dillane D, Sessler DI, Sieber F, Magaziner J, Marcantonio ER, Mehta S, Menio D, Ayad S, Stone T, Papp S, Schwenk ES, Elkassabany N, Marshall M, Jaffe JD, Luke C, Sharma B, Azim S, Hymes RA, Chin KJ, Sheppard R, Perlman B, Sappenfield J, Hauck E, Hoeft MA, Giska M, Ranganath Y, Tedore T, Choi S, Li J, Kwofie MK, Nader A, Sanders RD, Allen BFS, Vlassakov K, Kates S, Fleisher LA, Dattilo J, Tierney A, Stephens-Shields AJ, Ellenberg SS; REGAIN Investigators. Spinal Anesthesia or General Anesthesia for Hip Surgery in Older Adults. N Engl J Med. 2021 Nov 25;385(22):2025-2035. doi: 10.1056/NEJMoa2113514. Epub 2021 Oct 9. PMID 34623788